CLINICAL TRIAL: NCT02841579
Title: A Phase IIa Clinical Trial to Evaluate the Safety and Efficacy of Osimertinib (AZD9291) in First-line Patients With EGFR Mutation-positive Locally Advanced or Metastatic NSCLC and Concomitant EGFR T790M Mutation at Time of Diagnosis
Brief Title: Osimertinib (AZD9291) in First-line Locally Advanced or Metastatic NSCLC Patients With EGFR and EGFR T790M
Acronym: AZENT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP112; 2015-004828-66 (EudraCT Number)
Record Dates: First submitted 2016-07-08; First posted 2016-07-22 (Estimated); Results first posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Osimertinib (Experimental): The patients will be treated with 1 tablet of osimertinib (AZD9291) 80 mg per os (p.o.) daily. Patients will receive study treatment until disease progression or occurrence of unacceptable side effects up to 78 weeks from the time of the first administered dose.
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — The patients will be treated with 1 tablet of osimertinib (AZD9291) 80 mg per os (p.o.) daily up to 78 weeks from the time of the first administered dose.
  Other Names: AZD9291

SUMMARY:
The primary goal is to evaluate the efficacy of osimertinib (AZD9291), in terms of the objective response rate in patients with advanced non-squamous NSCLC with EGFR mutations and the EGFR T790M mutation at diagnosis as defined by RECIST 1.1 criteria.

Safety and efficacy will also be measured.

DETAILED DESCRIPTION:
Naïve patients ≥ 18 years of age with histological confirmation of locally advanced or metastatic, non-squamous non-small cell lung cancer (NSCLC) with an activating EGFR mutation and concomitant T790M mutation. Evidence of measurable or evaluable metastatic disease is required.

Primary objective:

* To evaluate the efficacy of osimertinib (AZD9291), in terms of the objective response rate in patients with advanced non-squamous NSCLC with EGFR mutations and the EGFR T790M mutation at diagnosis as defined by RECIST 1.1 criteria.

Secondary objectives:

* To determine the safety and tolerability profile of osimertinib (AZD9291), measured using the number and severity of AEs entered into the Case Report Form (CRF); chemistry, blood count, vital signs, physical examination, weight, ECG and performance status (S).
* To determine other efficacy parameters such as progression-free survival (PFS), overall survival (OS), time to treatment failure (TTF), duration of response (DOR), disease control rate (DCR), and tumor shrinkage (TS).
* To correlate the parameters of clinical response efficacy documented with the EGFR mutational status.
* To carry out a longitudinal analysis of EGFR mutations (including the T790M mutation) in plasma and serum.
* To determine levels of BIM mRNA as well as mRNA levels of other biomarkers related to EGFR TKI response and determine whether they are predictors of treatment response.
* To identify mechanisms of acquired resistance to osimertinib (AZD9291); mutations at the site of covalent binding to the drug (C797) or other mutations in tissue or blood.

Type of study: Multicenter, international, single-arm, open-label, non-controlled phase IIa clinical study.

Treatment: Patients will be treated with 1 tablet of osimertinib (AZD9291) 80 mg per os (p.o.) daily.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Patients with histological confirmation of locally advanced or metastatic, non-squamous non-small cell lung cancer (NSCLC) with an activating EGFR mutation and concomitant T790M mutation who are not candidates for local curative treatment.
* Patients with a M1a stage according to the TNM version 7 including M1a (malignant effusion) or M1b (distant metastasis), or locally advanced disease that is not a candidate for curative treatment (including patients who progress after chemoradiotherapy in stage III disease).
* Patients with a EGFR deletion or mutation in exon 19, exon 21 (L858R, L861Q) or exon 18 (G719X) and concomitant T790M mutation before treatment confirmed centrally.
* ECOG (Eastern Cooperative Oncology Group) performance status less than or equal to 2.
* Existence of measurable or evaluable disease (as per RECIST 1.1 criteria). Patients with asymptomatic and stable brain metastases are eligible for the study.
* Possibility of obtaining sufficient tissue sample, via a biopsy or surgical resection of the primary tumor or metastatic tumor tissue, within the 60 days prior to study entry.
* Life expectancy ≥12 weeks.
* Adequate hematologic function:

  * Absolute neutrophil count (ANC) > 1.5 x 109/L
  * platelet count > 100.0 x109/L
  * hemoglobin > 9.0 g/dL (> 6.2 mmol/L).
* Adequate coagulation: INR ≤ 1.5.
* Adequate liver function
* Adequate renal function.
* Capacity to swallow, patient capable of completing treatment and accessible, ensuring proper follow-up.
* Patients able to complete study and within geographical proximity allowing for adequate follow-up.
* Resolution of all acute toxic effects of previous anti-cancer therapy (which can only be adjuvant or neoadjuvant) or surgical interventions not exceeding grade ≤ 1 according to the NCI CTCAE version 4.0 (except for alopecia or other side effects that the investigator does not consider to be a risk to patient safety).
* All men or women of childbearing potential must use a contraception method during the study treatment and for at least 12 months after the last dose of the study drug.
* Signed and dated informed consent form

Exclusion Criteria:

* Locally advanced lung cancer candidate for curative treatment through radical surgery and/or radio(chemo)therapy.
* Patients diagnosed with another lung cancer subtype, patients with mixed NSCLC with predominantly squamous cell cancer, or with any small-cell lung cancer component.
* Patients with a EGFR deletion or mutation in exon 19, exon 21 (L858R, L861Q) or exon 18 (G719X) and concomitant T790M mutation before treatment that have not been confirmed centrally.
* Patients who have received prior antineoplastic treatment for advanced disease.
* Second active neoplasia
* Patients with just one measurable or evaluable tumor lesion that has been resected or irradiated prior to their enrollment in the study.
* Medical history of Interstitial Lung Disease (ILD) induced by drugs, radiation pneumonitis requiring steroid treatment or any evidence of clinically active ILD.
* Corrected QT Interval (QTc) >470 msec, obtained from 3 ECGs at rest, using the QTc value determined according to the clinical screening ECG machine.
* Any clinically significant abnormality in ECG rhythm, conduction or morphology at rest.
* Any factor that increases the risk of QTc prolongation or risk of irregular heartbeat or sudden inexplicable death under the age of 40 in first-degree relatives or any concomitant medications that prolong the QT interval.
* Uncontrolled, active or symptomatic metastases of CNS, carcinomatous meningitis or leptomeningeal disease indicated by known clinical symptoms, cerebral edema and/or progressive neoplasia. Patients with history of CNS metastasis or compression of the spinal cord are eligible if they have received local final treatment (e.g., radiotherapy, stereotactic surgery) and if they have remained clinically stable without using anticonvulsants and corticosteroids for a minimum of 4 weeks prior to the first day of study treatment.
* Refractory nauseas and vomiting, chronic gastrointestinal disease, inability to swallow study drug or significant intestinal resection that restricts the adequate absorption of osimertinib (AZD9291).
* Patients who have had a surgical procedure unrelated to the study within 7 days prior to the administration of the drug or a significant traumatic lesion during the 4 weeks prior to starting the administration of the study drug, patients who have not recovered from the side effects of any major surgery or patients who might need major surgery during the course of the study.
* Pregnant or breastfeeding women. Women of childbearing potential, including women who had their last menstrual period within the last two years, must have a negative serum or urine pregnancy test in the 7 days prior to the start of the treatment.
* Patients who are not willing to use an adequate contraception method until 12 months after the last dose of study treatment.
* Patients with a serious concomitant systemic disorder (e.g., active infection, including HIV or heart disease) that is incompatible with the study (in the opinion of the investigator), history of bleeding diathesis or anticoagulant therapy (the use of low molecular weight heparin is permitted provided that it is used for prophylaxis).
* Patients with a history of cancer that has been completely treated, with no evidence of malignant disease currently cannot be enrolled in the study if their chemotherapy was completed less than 6 months prior and/or have received a bone marrow transplant less than 2 years before the first day of study treatment.
* Prior treatment with cytotoxic chemotherapy for advanced NSCLC; neoadjuvant/adjuvant chemotherapy is permitted if at least 6 months have elapsed between the end of chemotherapy and the first day of study treatment.
* Patients who have received prior EGFR treatments for lung cancer.
* Patients who have received treatment with an investigational drug within 3 weeks before the first day of study treatment.
* Treatment with prohibited drugs within 14 days before the first day of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-09-02 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2020-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Rosell, MD, PhD, Principal Investigator — Catalan Institute of Oncology, Institut d'Investigació en Ciències de la Salut Germans Trias i Pujol
Locations (6):
- Spain (6):
  - MedSIR Investigative Site, A Coruña
  - MedSIR Investigative Site, Barcelona
  - MedSIR Investigative Site, Bilbao
  - MedSIR Investigative Site, Madrid
  - MedSIR Investigative Site, Málaga
  - MedSIR Investigative Site, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Majem M, Sullivan I, Viteri S, Lopez-Vivanco G, Cobo M, Sanchez JM, Garcia-Gonzalez J, Garde J, Sampayo M, Martrat G, Malfettone A, Karachaliou N, Molina-Vila MA, Rosell R. First-line osimertinib in patients with epidermal growth factor receptor-mutant non-small-cell lung cancer and with a coexisting low allelic fraction of Thr790Met. Eur J Cancer. 2021 Dec;159:174-181. doi: 10.1016/j.ejca.2021.09.039. Epub 2021 Nov 8. PMID 34763195

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Fifty-one patients were screened of whom 22 patients with advanced NSCLC harbouring pre-treatment sensitising EGFR and Thr790Met mutations were enrolled and started to receive first-line osimertinib.
Period: Overall Study
Arm/Group | Osimertinib
Started | 22
Completed | 11
Not Completed | 11
Not completed — Death | 1
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 9

BASELINE CHARACTERISTICS:
Arm/Group | Osimertinib
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 21
  Black | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 22
Smoking history [Count of Participants; unit: Participants]
  Never | 13
  Former | 9
Tumor stage [Count of Participants; unit: Participants] — Tumor stage was assessed at baseline according to TNM classification version 7, in which higher grades are correlated with worse outcomes.
  Participants
    IIIB | 2
    IV | 20
Central nervous system metastases [Count of Participants; unit: Participants]
  Yes | 3
  No | 19
EGFR sensitizing mutation [Count of Participants; unit: Participants] — EGFR mutation testing was determined in tissue and blood samples using a Taqman assay. For sensitizing mutations, a tissue sample was considered positive if the two cell extracts collected were positive. In blood samples, analyses were performed using two samples of serum and/or two samples of plasma cfDNA per patient.
  Participants
    Ex19del | 6
    Thr790Met | 2
    Leu858Arg | 8
Tissue EGFR sensitizing mutation [Count of Participants; unit: Participants] — EGFR mutation testing was determined in tissue samples using a Taqman assay. For sensitizing mutations, a tissue sample was considered positive if the two cell extracts collected were positive.
  Participants
    Gly719X | 3
    Ex19del | 10
    Thr790Met | 22
    Leu858Arg | 9

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Defined as the percentage of patients who achieved complete response [CR] and partial response [PR] to treatment in accordance to the revised RECIST guidelines (version 1.1) for target lesions: CR, disappearance of all target lesions; PR: at least 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Through study completion. From baseline up to approximately 28 months.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Osimertinib
Number analyzed (Participants) | 22
percentage of patients | 77.3 [54.6 to 89.3]

2. Secondary Outcome: Overall Survival (OS)
Description: Time from the start of treatment to the time of death due to any cause.
Time Frame: Through study completion. From baseline up to 41 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Osimertinib
Number analyzed (Participants) | 22
months | 28.39 [25.62 to NA] — The median survival of 28.39 months was reached during the study; however, the upper limit of the confidence interval is not available due to an insufficient number of participants with events beyond the median value. Patients who had not experienced the event were censored at their last known follow-up date. This limitation arises because the calculation of the upper limit requires a sufficient number of events after the median, which was not the case in this study.

3. Secondary Outcome: Duration of Response (DoR)
Description: Time from the first documented response to documented disease progression or death, in accordance with RECIST 1.1 criteria.
Time Frame: Through study completion. From baseline up to 41 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Osimertinib
Number analyzed (Participants) | 22
months | 20.0 [11.2 to NA] — The upper limit of the confidence interval for the median Duration of Response (DoR) could not be determined due to an insufficient number of participants with events beyond the observed median.

4. Secondary Outcome: Disease Control Rate
Description: Percentage of patients with complete response, partial response or stable disease for a minimum of 24 weeks, assessed in accordance with the modified Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1, during all study period from baseline up to 78 weeks from the time of the first administration dose
Time Frame: Through study completion. From baseline up to 41 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib
Number analyzed (Participants) | 22
Participants | 19

5. Secondary Outcome: Tumor Shrinkage
Description: Number of patients that presented tumor shrinkage
Time Frame: Through study completion. From baseline up to 41 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib
Number analyzed (Participants) | 22
Participants | 17

6. Secondary Outcome: Overall Plasma EGFR Mutation Status at Baseline
Description: Percentage of patients with a positive sensitizing EGFR mutation in plasma at baseline
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib
Number analyzed (Participants) | 21
Participants | 15

7. Secondary Outcome: Overall Plasma Acquired Resistance to Osimertinib (AZD9291)
Description: Percentage of patients who develop anti-drug mutations in plasma
Time Frame: Through study completion. From baseline up to 41 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib
Number analyzed (Participants) | 12
Participants | 7

8. Secondary Outcome: Number of Participants With Grade 3 or 4 Adverse Events and SAEs
Description: Patient safety and adverse events will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) of the U.S. National Cancer Institute (NCI), version 4. Adverse event(s) are those which, according to the protocol or in the opinion of the investigator, can cause serious or permanent damage or which rule out further treatment with the study drug. Grade 3 means severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 means life-threatening consequences; urgent intervention indicated.
Time Frame: Through study completion. From baseline up to 41 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib
Number analyzed (Participants) | 22
Participants | 10

9. Secondary Outcome: Progression-free Survival
Description: Defined as the period of time from treatment initiation to the first occurrence of disease progression or death from any cause, whichever occurs first, as determined locally by the investigator using RECIST v.1.1.
Time Frame: Through study completion. From baseline up to 41 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Osimertinib
Number analyzed (Participants) | 22
months | 23.1 [14.1 to NA] — The median progression-free survival (PFS) was 23.1 months; however, the upper limit of the confidence interval is not available due to an insufficient number of participants who experienced disease progression or death beyond the median value. Patients who had not progressed or died at the time of analysis were censored at their last evaluable assessment.

10. Secondary Outcome: Overall Plasma EGFR Mutation Status at Two Weeks After the First Study Dose
Description: Measured by percentage of patients with a positive sensitizing EGFR mutation in plasma two weeks after the first study dose
Time Frame: Two weeks after the first study dose
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib
Number analyzed (Participants) | 21
Participants | 5

11. Secondary Outcome: Overall Plasma EGFR Mutation Status at Disease Progression
Description: Measured by percentage of patients with a positive sensitizing EGFR mutation in plasma at disease progression
Time Frame: At the time of disease progression confirmed radiologically or clinically, up to 78 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib
Number analyzed (Participants) | 12
Participants | 8

12. Secondary Outcome: Plasma EGFR Thr790Met Mutation Status at Baseline
Description: Measured by percentage of patients with EGFR Thr790Met mutation in plasma at baseline
Time Frame: At baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib
Number analyzed (Participants) | 21
Participants | 2

13. Secondary Outcome: Plasma EGFR Thr790Met Mutation Status at Two Weeks After the First Study Dose
Description: Measured by percentage of patients with EGFR Thr790Met mutation in plasma at two weeks after the first study dose
Time Frame: Two weeks after the first study dose
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib
Number analyzed (Participants) | 21
Participants | 2

14. Secondary Outcome: Plasma EGFR Thr790Met Mutation Status at Disease Progression
Description: Measured by percentage of patients with EGFR Thr790Met mutation in plasma at disease progression
Time Frame: At the time of disease progression confirmed radiologically or clinically, up to 78 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib
Number analyzed (Participants) | 12
Participants | 2

ADVERSE EVENTS:
Time Frame: 42 months
Description: Regular investigator and local laboratory assessments were used to determine adverse events. Basic safety visits were performed on day 1 of each cycle every 2 cycles (every 6 weeks).
Arm/Group | Osimertinib
All-Cause Mortality (participants affected / at risk) | 1/22
Serious Adverse Events (participants affected / at risk) | 10/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Osimertinib (N=22)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Atrioventricular block (Cardiac disorders) | 1
Elevated creatine phosphokinase levels in blood (Musculoskeletal and connective tissue disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Limb pain (Musculoskeletal and connective tissue disorders) | 1
Disease worsening (General disorders) | 1
Femur fracture (Musculoskeletal and connective tissue disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1
Paralytic ileus (Gastrointestinal disorders) | 1
Pulmonary infection (Infections and infestations) | 1
Heart failure (Cardiac disorders) | 1
Peripheral ischemia (Vascular disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Psychotic disorders (Psychiatric disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Osimertinib (N=22)
Diarrhoea (Gastrointestinal disorders) | 17
Asthenia (General disorders) | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Constipation (Gastrointestinal disorders) | 7
Anorexia (General disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
Respiratory tract infection (Infections and infestations) | 5
Alopecia (General disorders) | 4
Dry mouth (Skin and subcutaneous tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 7
Mucosa inflammation (Immune system disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 3
Muscle spasm (Musculoskeletal and connective tissue disorders) | 3
Upper respiratory tract infection (Infections and infestations) | 3
Insomnia (General disorders) | 3
Dizziness (General disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 6
Itching (Skin and subcutaneous tissue disorders) | 3
Dry nose (Skin and subcutaneous tissue disorders) | 3
Ungual toxicity (Skin and subcutaneous tissue disorders) | 3
Sensory disturbances (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Cold (Infections and infestations) | 2
Headache (Nervous system disorders) | 2
Congested nose (Infections and infestations) | 2
Exertional dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Edema (General disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Deep vein thrombosis (Vascular disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Gastroenteritis (Infections and infestations) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2
Urinary tract infections (Infections and infestations) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Nasopharyngitis (Infections and infestations) | 2
Nausea (Gastrointestinal disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Paronychia (Infections and infestations) | 2
Elevated transaminase levels (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT02841579/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT02841579/SAP_001.pdf